CLINICAL TRIAL: NCT00950014
Title: Testing Numeric Formats for Presenting Data About Treatment Benefits and Harms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Attorney General Consumer & Prescriber Education Grant (Other)
Responsible Party: Lisa M. Schwartz, MD, MS, White River Junction VAMC
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 16783
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2009-07

CONDITIONS: Risk Communication
Keywords: Numeracy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Percentage format only (Experimental): Numbers are presented in percentage format (e.g., 35%, 0.2%) only.
  Interventions: Other: Presentation of drug efficacy and side effect data
- Fixed frequency format only (Experimental): Numbers are presented in fixed frequency format only (5 out of 1000, 0.6 out of 1000). Denominators remains the same for each number.
  Interventions: Other: Presentation of drug efficacy and side effect data
- Variable frequency format (Experimental): Frequency denominators are adjusted to keep the numerator greater than 1, so they may change throughout the survey (e.g., 6 out of 1000, 42 out of 100)
  Interventions: Other: Presentation of drug efficacy and side effect data
- Fixed combination format (Active Comparator): Numbers are presented with both percentages and frequencies, and frequency denominators remain fixed (e.g., _ out of 1000).
  Interventions: Other: Presentation of drug efficacy and side effect data
- Variable combination format (Experimental): Numbers are presented with both percentages and frequencies, but frequency denominators may vary (e.g., _ out of 1000, _ out of 100).
  Interventions: Other: Presentation of drug efficacy and side effect data

INTERVENTIONS:
Other: Presentation of drug efficacy and side effect data — Data presented in 1 of 5 numeric formats in each arm: percentage only, fixed frequency only, variable frequency, variable combination and fixed combination format.

SUMMARY:
The purpose of this study is to test comprehension of five numeric formats used to present data about treatment benefits and harms.

ELIGIBILITY:
Inclusion criteria

* Participants will be randomly selected from a research panel of more than 60,000 U.S. households (Knowledge Networks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2944 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Comprehension questions (e.g., overall direction of effect and specific numeric data) | 0 weeks (assessed during intervention)

SECONDARY OUTCOMES:
Risk perceptions (e.g., how big or small is the benefit)and preferences (e.g., did the box help subjects understand the benefits) assessed via Internet surveys. | 0 weeks (assessed during intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Schwartz, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center; Steven Woloshin, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center

REFERENCES:
- [Background] Schwartz LM, Woloshin S, Welch HG. Using a drug facts box to communicate drug benefits and harms: two randomized trials. Ann Intern Med. 2009 Apr 21;150(8):516-27. doi: 10.7326/0003-4819-150-8-200904210-00106. Epub 2009 Feb 16. PMID 19221371
- [Background] Schwartz LM, Woloshin S, Welch HG. The drug facts box: providing consumers with simple tabular data on drug benefit and harm. Med Decis Making. 2007 Sep-Oct;27(5):655-62. doi: 10.1177/0272989X07306786. Epub 2007 Sep 14. PMID 17873258
- [Derived] Woloshin S, Schwartz LM. Communicating data about the benefits and harms of treatment: a randomized trial. Ann Intern Med. 2011 Jul 19;155(2):87-96. doi: 10.7326/0003-4819-155-2-201107190-00004. PMID 21768582